CLINICAL TRIAL: NCT00783484
Title: A Double-Blind (3rd Party Open), Placebo-Controlled, Crossover, Dose Escalating Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Single Oral Doses Of PF-03716539, To Assess The Potential Of PF-03716539 To Inhibit CYP3A4 (In Vivo) And To Evaluate The Drug Interaction Potential Between PF-03716539 And Darunavir Or Maraviroc In Healthy Adult Subjects
Brief Title: A Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Single Oral Doses Of PF-03716539 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B0831001
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Volunteers
Keywords: First in Human (FIH), PF-03716539, PK enhancer
MeSH Terms: interventions — Midazolam; Darunavir; Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): PF-03716539 crossover, single dose escalation (doses subject to change).
  Interventions: Drug: PF-03716539; Other: Placebo
- Cohort 2 (Experimental): PF-03716539 crossover, single dose escalation (doses subject to change).
  Interventions: Drug: PF-03716539; Other: Placebo
- Cohort 3 (Experimental): Midazolam-PF-03716539 drug-drug interaction (PF-03716539 doses subject to change).
  Interventions: Drug: Midazolam; Drug: Midazolam + PF-03716539 (100 mg); Drug: Midazolam + PF-03716539 (50 mg)
- Cohort 4 (Experimental): Darunavir-PF-03716539 drug-drug interaction (PF-03716539 doses subject to change).
  Interventions: Drug: Darunavir; Drug: Darunavir + PF-03716539
- Cohort 5 (Experimental): Maraviroc-PF-03716539 drug-drug interaction (PF-03716539 doses subject to change).
  Interventions: Drug: Maraviroc; Drug: Maraviroc +PF-03716539
- Cohort 6 (Experimental): Maraviroc-PF-03716539 drug-drug interaction (PF-03716539 200 mg).
  Interventions: Drug: Maraviroc; Drug: Maraviroc +PF-03716539

INTERVENTIONS:
Drug: PF-03716539 — PF-03716539 10 mg oral solution, single dose
  Arms: Cohort 1
Drug: PF-03716539 — PF-03716539 25 mg oral solution, single dose
  Arms: Cohort 1
Drug: PF-03716539 — PF-03716539 3 mg oral solution, single dose
  Arms: Cohort 1
Other: Placebo — Placebo for 3 mg, 10 mg and 25 mg of PF-03716539 (single dose)
  Arms: Cohort 1
Drug: PF-03716539 — PF-03716539 100 mg oral solution, single dose
  Arms: Cohort 2
Drug: PF-03716539 — PF-03716539 200 mg oral solution, single dose
  Arms: Cohort 2
Drug: PF-03716539 — PF-03716539 50 mg oral solution, single dose
  Arms: Cohort 2
Other: Placebo — Placebo for 50 mg, 100 mg and 200 mg of PF-03716539 (single dose)
  Arms: Cohort 2
Drug: Midazolam — Midazolam 1 mg IV, single dose
  Arms: Cohort 3
Drug: Midazolam + PF-03716539 (100 mg) — Midazolam 1 mg IV, single dose plus PF-03716539 100 mg oral solution, single dose
  Arms: Cohort 3
Drug: Midazolam + PF-03716539 (50 mg) — Midazolam 1 mg IV, single dose plus PF-03716539 50 mg oral solution, single dose
  Arms: Cohort 3
Drug: Darunavir — Darunavir 600 mg tablet twice daily for 9 days (Days 1-9)
  Arms: Cohort 4
Drug: Darunavir + PF-03716539 — Darunavir 600 mg tablet, single dose plus PF-03716539 50 mg oral solution, single dose (Day 10)
  Arms: Cohort 4
Drug: Maraviroc — Maraviroc 150 mg tablet once daily for 6 days (Days 1-6)
  Other Names: Selzentry
  Arms: Cohort 5
Drug: Maraviroc +PF-03716539 — Maraviroc 150 mg tablet, single dose plus PF-03716539 100 mg oral solution, single dose (Day 7)
  Other Names: Selzentry
  Arms: Cohort 5
Drug: Maraviroc — Maraviroc 225 mg tablet once daily for 6 days (Days 1-6)
  Other Names: Selzentry
  Arms: Cohort 6
Drug: Maraviroc +PF-03716539 — Maraviroc 225 mg tablet, single dose plus PF-03716539 200 mg oral solution, single dose (Day 7)
  Other Names: Selzentry
  Arms: Cohort 6

SUMMARY:
First in human study to evaluate the safety, tolerability, and pharmacokinetics of PF-03716539. The potential of PF-03716539 to increase the concentrations of midazolam, darunavir and maraviroc will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.

Body Mass Index (BMI) of approximately 18 to 30 kg/m2. Total body weight >50 kg (110 lbs).

Exclusion Criteria:

Pregnant or nursing females. females of childbearing potential. Evidence or history of clinically significant hematological, renal (including kidney stones), endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or clinical findings at screening.

Treatment with an investigational drug within 30 days (or determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of escalating single oral doses of PF 03716539 administered as Extemporaneous Powder for Solution (EPS) in healthy adult subjects. | 27 days
To explore the pharmacokinetics of escalating single oral doses of PF 03716539 in healthy adult subjects. | 6 days

SECONDARY OUTCOMES:
To assess the potency of PF 03716539 for CYP3A4 inhibition utilizing single dose IV midazolam as a probe substrate for CYP3A4/5. | 6 days
To evaluate the potential of PF 03716539 to enhance or "boost" the pharmacokinetics of both darunavir and maraviroc. | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0831001&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20Single%20Oral%20Doses%20Of%20PF-03716539%20In%20Healthy%20Adult%20Subjects